# The Effect of Tranexamic Acid on Calculated Total Blood Loss in Patients undergoing Revision Shoulder Arthroplasty

This is a phase IV, randomized, single-blind, single-center study comparing calculated total blood loss, surgical drain output and hematoma formation in patients who receive 2 doses of Tranexamic Acid (TXA) versus control group undergoing revision total shoulder arthroplasty. Patients will be randomized to either receive 2 doses of IV TXA, first dose prior to surgical incision and second dose given 3 hours later or to the *control group*, where no TXA will be administered.

| Principal Investigator: | Principal Investigator: Arthur C. Hertling, MD, MBA |
|---|---|
| | Department of Anesthesiology, Perioperative Care and Pain Med |
| | NYU Langone Health |
| | NYU Langone Orthopedic Hospital |
| | 301 East 17 <sup>th</sup> Street |
| | New York, NY 10003 |
| | Arthur.Hertling@nyulangone.org |
| | O: (212) 598-6085 |
| Additional Investigators: | |
| Table 1 Color Co | Young Kwon, MD, PhD |
| | Department of Orthopedic Surgery |
| | NYU Langone Health |
| | NYU Langone Orthopedic Hospital |
| | 301 East 17 <sup>th</sup> Street |
| | New York, NY 10003 |
| | Young.Kwon@nyulangone.orgO:(646) 501-7170 |
| | Mandeep Virk, MD |
| | Department of Orthopedic Surgery |
| | Department of Orthopedic Surgery |
| | NYU Langone Health |
| | NYU Langone Orthopedic Hospital |
| | 301 East 17 <sup>th</sup> Street |
| | New York, NY 10003 |
| | Mandeep.Virk@nyulangone.org |
| | O: (646) 754-2100 |
| | Jasanh Zuakarman MD |
| | Joseph Zuckerman, MD |
| | Department of Orthopedic Surgery |
| | NYU Langone Health |
| | NYU Langone Orthopedic Hospital |
| | 301 East 17 <sup>th</sup> Street |
| | New York, NY 10003 |
| | Joseph.Zuckerman@nyulangone.org |
| | O: (212) 598-6674 |
| | CONFIDENTIAL |

Page 2

| Devisions with the distant. | Page 2 |
|---|---|
| | Jesse Ng, MD |
| | Department of Anesthesiology, Perioperative Care and Pain Med |
| | NYU Langone Health NYU Langone Orthopedic Hospital 301 East 17 <sup>th</sup> Street New York, NY 10003 Jesse.Ng@nyulangone.org O: (212) 598-6085 |
| | Germaine Cuff, PhD Department of Anesthesiology, Perioperative Care and Pain Med |
| | NYU Langone Health<br>NYU Tisch Hospital<br>550 1st Ave |
| | New York, NY 10016 Germaine.Cuff@nyulangone.org O: (212) 263-5072 |
| NYULMC Study Number: | S20-01617 |
| Study Product: | |
| ClinicalTrials.gov Number | |

**Initial version:** 11/20/2020 **Amended:** 05/05/2022

Amended:

Version: 1.0 dated 05/05/2022

### **Statement of Compliance**

This study will be conducted in accordance with the Code of Federal Regulations on the Protection of Human Subjects (45 CFR Part 46), 21 CFR Parts 50, 56, 312, and 812 as applicable, any other applicable US government research regulations, and institutional research policies and procedures. The International Conference on Harmonisation ("ICH") Guideline for Good Clinical Practice ("GCP") (sometimes referred to as "ICH-GCP" or "E6") will be applied only to the extent that it is compatible with FDA and DHHS regulations. The Principal Investigator will assure that no deviation from, or changes to the protocol will take place without prior agreement from the sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants. All personnel involved in the conduct of this study have completed Human Subjects Protection Training.

Study number: S20-01617 Version: 1.0 dated 05/05/2022

# **Table of Contents**

| $\mathbf{S}'$ | STATEMENT OF COMPLIANCE | |
|---|---|---|
| L | IST OF ABBREVIATIONS | t |
| | ROTOCOL SUMMARY | |
| | KEY ROLES | |
| 1 | | |
| 2 | BACKGROUND AND SPECIFIC AIMS | 8 |
| | 2.1 Specific Aims | |
| | 2.1 STATISTICAL HYPOTHESES | |
| | 2.2 OBJECTIVES AND PURPOSE | |
| 3 | STUDY DESIGN AND ENDPOINTS | 10 |
| | 3.1 DESCRIPTION OF STUDY DESIGN | 10 |
| | 3.2 SCHEMATIC OF STUDY DESIGN | 11 |
| 4 | STUDY ENROLLMENT AND WITHDRAWAL | 12 |
| | 4.1 Inclusion Criteria | 10 |
| | 4.2 EXCLUSION CRITERIA | |
| | 4.3 VULNERABLE SUBJECTS | |
| | 4.4 RECRUITMENT AND CONSENT | 12 |
| | 4.5 DURATION OF STUDY PARTICIPATION | |
| | 4.6 TOTAL NUMBER OF PARTICIPANTS AND SITES | |
| | 4.7 PARTICIPANT WITHDRAWAL OR TERMINATION | |
| | 4.8 Premature Termination or Suspension of Study | |
| 5 | RISKS AND BENEFITS | 14 |
| | 5.1 POTENTIAL RISKS | 14 |
| | 5.2 POTENTIAL BENEFITS | 14 |
| 6 | STATISTICAL ANALYSIS | 17 |
| | 6.1 GENERAL APPROACH | 17 |
| | 6.2 ANALYSIS OF ENDPOINTS | |
| | 6.2.1 Baseline Descriptive Statistics | 18 |
| | 6.3 SAMPLE SIZE | |
| | 6.4 ENROLLMENT/RANDOMIZATION/MASKING PROCEDURES | |
| | 6.5 Breaking the Study Blind/Participant Code | |
| 7 | ASSESSMENT OF SAFETY | 18 |
| | 7.1 DEFINITION OF SERIOUS ADVERSE EVENTS (SAE) | 18 |
| | 7.2 CLASSIFICATION OF AN ADVERSE EVENT | |
| | 7.2.1 Severity of Event | |
| | 7.2.2 Relationship to Study Agent | |
| | 7.3 TIME PERIOD AND FREQUENCY FOR EVENT ASSESSMENT AND FOLLOW-UP | |
| | 7.4 SAFETY OVERSIGHT | |
| 8 | SOURCE DOCUMENTS AND ACCESS TO SOURCE DATA/DOCUMENTS | 21 |
| 9 | ETHICS/PROTECTION OF HUMAN SUBJECTS | 27 |

Page 5

Study number: S20-01617 Version: 1.0 dated 05/05/2022

| 9.1 | ETHICAL STANDARD | 22 |
|-------|-------------------------------------------------|----|
| 9.2 | INSTITUTIONAL REVIEW BOARD | 22 |
| 9.3 | PARTICIPANT AND DATA CONFIDENTIALITY | 22 |
| 10 DA | TA HANDLING AND RECORD KEEPING | 23 |
| 10.1 | DATA COLLECTION AND MANAGEMENT RESPONSIBILITIES | 23 |
| 10.2 | STUDY RECORDS RETENTION | 23 |
| 10.3 | PROTOCOL DEVIATIONS | 23 |
| 10.4 | PUBLICATION AND DATA SHARING POLICY | 23 |
| 11 ST | UDY FINANCES | 24 |
| 11.1 | FUNDING SOURCE | 24 |
| 11.2 | COSTS TO THE PARTICIPANT | |
| 11.3 | PARTICIPANT REIMBURSEMENTS OR PAYMENTS | 24 |
| 12 CO | NFLICT OF INTEREST POLICY | 24 |
| 13 RE | FERENCES | 25 |
| 14 AT | TACHMENTS | 25 |

Study number: S20-01617 Page 6 Version: 1.0 dated 05/05/2022

### **List of Abbreviations**

AE Adverse event

ANOVA Analysis of variance; a linear model

ASA American Society of Anesthesiologist Score

CI Confidence interval

DVT Deep vein thrombosis

IV Intravenous

MI Myocardial Infarction

NSAID Non-steroidal anti-inflammatory drug

PACU Post-Anesthesia Care Unit

PE Pulmonary Embolus

PO Taken orally

PRN Taken as needed

Q4h Taken every four hours

SAE Serious adverse event

SD Standard deviation; a parameter that characterizes a population distribution

SE Standard error

TID Taken three times per day

TSA Total Shoulder Arthroplasty

TXA Tranexamic Acid

VAS Visual analog scale

Study number: S20-01617 Page 7 Version: 1.0 dated 05/05/2022

# **Protocol Summary**

| 1 Totocoi Sullillai y | |
|---|---|
| Title | The Effect of Tranexamic Acid in Patients undergoing Revision Total<br>Shoulder Athroplasty |
| Short Title | TXA in Revision Total Shoulder Arthroplasty |
| Brief Summary | This is a phase IV, randomized, single-blind, single-center study comparing calculated total blood loss, surgical drain output and hematoma formation in patients who receive 2 doses of Tranexamic Acid (TXA) versus control group undergoing revision total shoulder arthroplasty. Patients will be randomized to either receive 2 doses of IV TXA, first dose prior to surgical incision and second dose given 3 hours later or to the <i>control group</i> , where no TXA will be administered. |
| Phase | Clinical study phase IV |
| Objectives | To compare the effectiveness of IV TXA on reducing calculated total blood loss, surgical drain output and hematoma formation in patients undergoing revision total shoulder arthroplasty. |
| Methodology | phase IV, randomized, single-blind, single-center study |
| Endpoints | Primary Endpoints: |
| Study Duration | 3 years |
| Participant Duration | 2 weeks |
| Population | 82 participants scheduled for Revision Total Shoulder Arthroplasty |
| Study Sites | NYU Langone Orthopedic Hospital (LOH) |
| Number of participants | 82 participants |
| Description of Study<br>Agent/Procedure | Injection of 1 gram of IV TXA before surgical plus 1 gram of IV TXA three hours later |
| Reference Therapy | Reference is No TXA (control) |
| Key Procedures | Injection of Tranexamic Acid |
| Statistical Analysis | Intention-to-treat analysis will be performed with mean, t-tests, within and between group ANOVA and linear regression, Wilcoxon's rank-sum |


### 1 Key Roles

### Principal Investigator:

### Arthur C. Hertling, MD, MBA

Department of Anesthesiology, Perioperative Care and Pain Med

NYU Langone Health NYU Langone Orthopedic Hospital 301 East 17<sup>th</sup> Street New York, NY 10003 <u>Arthur.Hertling@nyulangone.org</u> O: (212) 598-6085

### **Co-Investigator:**

### Young Kwon, MD, PhD

Associate Professor of Orthopedic Surgery Department of Orthopedic Surgery Center for Musculoskeletal Care NYU Langone Health 333 East 38<sup>th</sup> street New York, NY 10016

### 2 Background and Specific Aims

Anatomic total shoulder arthroplasty (TSA) and Reverse total shoulder arthroplasty (rTSA) are surgical procedures where the damaged glenohumeral joint is replaced by a metal and plastic prosthesis. This surgery is indicated to alleviate pain and treat rotator cuff tear arthropathy. The number of total shoulder arthroplasties has increased tremendously over the last ten years. With more than 53,000 shoulder replacement surgery done yearly in the US, (Agency for Healthcare Research and Quality) revision shoulder surgery is an inevitable consequence. Revision rates have been reported to be approximately 11% for hemi-arthroplasty and total anatomical implants, and 10% for reversed implants (Favard). Pain and shoulder pathology are indications for revision shoulder surgery. Failure is classified as soft-tissue deficiencies, osseous deficiencies, component wear, or infection (Dines). It is well known that perioperative blood loss after TSA is significant with blood transfusion rates varying from 4.5-43%. Included in the common risk factors are preoperative anemia, comorbities, and revision total shoulder surgery (Burns). Additional studies have shown that revision total shoulder arthroplaties have a rate of blood transfusion of 21-31% (King, Bryan).

Given the need to reduce perioperative blood loss and minimize transfusion risks, many clinicians use Tranexamic acid (TXA) to reduce orthopedic surgical complications. TXA is a synthetic lysine analog that inhibits the conversion of plasmin from plasminogen thereby preventing the breakdown of fibrin (McCormack). This action stabilizes blood clots and has been shown to decrease the risk of blood loss for several different types of orthopedic surgeries. TXA is increasingly used in orthopedic joint reconstructive surgery and has proven to be safe and effective in reducing blood loss following total knee arthroplasty (TKA) and total hip arthroplasty (THA) (Fillingham, Yang). More recently, it has been shown to reduce postoperative blood loss following primary total shoulder arthroplasty Kirsch).


There is clear evidence that TXA is beneficial in THA, TKA, and primary TSA. Currently, there is no data on whether TXA will reduce blood loss in patients undergoing revision TSA. We propose this randomized control study comparing intravenous versus control (i.e., no TXA) in hopes to define the benefit of TXA in patients undergoing revision total shoulder surgery.

The only FDA approved usage for TXA is for heavy menstrual bleeding and short term bleeding prevention in patients with hemophilia. TXA has been widely used off label to reduce blood loss in a variety of surgical cases. In orthropedics, TXA is commonly used in major spine surgery and total joint arthroplasty procedures. The benefit of TXA in reducing total blood loss and post operative transfusion in this population has been well supported in the literature (Budge, Kuo, Fillingham, Cvetanovich).

TXA is lawfully marketed and this investigation is not intended to be reported to FDA as a well-controlled study in support of a new indication for use nor intended to be used to support any other significant change in the labeling for the drug. This investigation does not involve a route of administration or dosage level or use in a patient population or other factor that significantly increases the risks (or decreases the acceptability of the risks) associated with the use of the drug product. TXA 1000mg will be administered to patients prior to incision and 3 hours after. This dose is standard practice at NYU Langone Orthopedic Hospital and no adverse events with TXA have been reported since the implementation of this dose and usage at our institution. Kirsch et al performed a systematic review and meta-analysis of the role of TXA in shoulder arthroplasty surgery. This review looked at a total of 629 patients enrolled in 5 studies. The dosing and route of administration of TXA varied among the studies (intravenously in 4 studies and topically in 1 study). The dosing of TXA varied for the studies the range included 10mg/kg bolus, 20mg/kg bolus or 1000mg bolus. For this meta-analysis, no thromboembolic events were associated with TXA use. (Kirsch) This investigation is conducted in compliance with the requirements for institutional review set forth in part 56 and with the requirements for informed consent set forth in part 50. This investigation is conducted in compliance with the requirements of 312.7 (re: promotion of investigational drugs

### 2.1 Specific Aims

**AIM:** To determine if the use of IV TXA results in a quantifiable decrease in perioperative calculated total blood loss and transfusion requirements in patients undergoing revision TSA.

### 2.2 Statistical Hypotheses

We hypothesize that patients who receive 2 doses of intravenous TXA will have a greater reduction in calculated total blood loss compared with patients who receive no TXA. Furthermore, intravenous TXA will be more effective in decreasing post op hematoma formation in comparison to the control group.

### **Objectives and Purpose**

The goal of this study is to compare the effectiveness of IV TXA vs control at reducing post-operative blood loss.

Primary outcomes measures will be calculated total blood loss and post op drain output, where the surgical drain output will be recorded by floor nurse every 8 hours in EPIC.

Secondary outcomes include formation of hematoma, need for blood transfusions and any other adverse events such development of DVT, PE, MI etc, that may occur.


# 3 Study Design and Endpoints

| Arm #1: IV TXA<br>(2 DOSES) | Arm #2: CONTROL<br>GROUP |
|---|---|
| Sample Size: 41 Subjects | Sample Size: 41 subjects |
| Medication: IV Tranxemic Acid | None (No TXA) |
| Total Dosage: 2 grams | N/A |
| 1 gram before surgical incision + 1 gram, 3 hours after first dose | |
| 1 gram, 3 nours after first dose | |

# 3.1 Description of Study Design

### PRE-SCREENING PHASE/CONSENTING PHASE:

Surgeons will inform eligible patients of the study during their pre-surgical visit in their office. Potential participants will be able to take the informed consent home to read through and take sufficient time to ask questions and/or discuss with family or research team prior to making an informed decision to participate. If the patient is agreeable, a member of the research team will provide further details and ask the patient to participate on day of surgery. An authorized research member will obtain informed consent prior to surgery.

### **RANDOMIZATION PHASE:**

Subjects scheduled to undergo revision TSA will be randomized to receive one of two treatment options. This study will utilize a simple randomization approach to generate two-equal groups. All subjects have an equal chance (1:2) of getting randomized into one of the two treatments groups: (1) Two doses of IV TXA, one before incision and the second 3 hours later. (2) control group – no TXA given. Randomization of each subject will be done on day of surgery. The randomization schedule will be generated using a computer software program such as randomization.com

### TREATMENT PHASE:

Subjects randomized to group 1 will receive an injection of 1 gram of IV TXA before surgical incision plus 1 gram of TXA IV 3 hours later. Subjects randmomized to group 2 will receive no TXA. Neither the anesthesiologist or surgeon will be blinded to the patient's group assignment, as they will be the one performing the treatment. All other stakeholders (patient, other caregivers, and research staff collecting the data) will be blinded to the patient's group assignment.

### **INTRA-OPERATIVE PHASE:**


As per standard practice at NYU Langone Orthopedic Hospital, all patients will receive an interscalene nerve block plus or minus general anesthesia. For the procedure, the surgeon will utilize a deltopectoral approach and use electrocautery for hemostasis throughout the procedure.

### Hemovac Drain:

Lastly, a single Hemovac drain will be placed at the end of the procedure, deep to the deltopectoral interval and will be removed prior to discharge on POD 1.

### **POST-OPERATIVE PHASE:**

The PACU nurse will administer the second dose of TXA for the patients who are in the second arm of TXA study, 3 hours after the first dose was administered.

### Hemoglobin Levels

On POD 1, the floor nurse will draw and send a post op hemoglobin/hematocrit panel for all study patients prior to discharge.

### Hemovac Surgical Output:

The floor nurse will also document the amount of blood in the indwelling hemovac surgical drain placed in the operative shoulder joint. The drain output will be documented every 8 hours in EPIC. We will record the drain output for the first 16 hours after surgery – essentially 2 output shifts. If patients are in the hospital longer, we will record the third 24 hour drain output.

### Hematoma:

As per standard practice, the Orthopedic resident or fellow will assess for the presence of hematoma on POD 1, prior to patient discharge. The surgeon will assess for presence of hematoma at the 2-week follow up visit. This information will be recorded in EPIC and the data will be used for the study.

### Total calculated blood loss:

The volume of perioperative blood loss will be determined on the basis of the blood volume and change in hemoglobin from preoperatively to 1 day postoperatively.

### **Blood Volume:**

Blood volume will be calculated using Nadler's formula. (Cventovich, Fillingham, Abildgard, Tsukada, Nadler) We will calculate the predicted blood volume of each patient according to the formula:

blood volume (L) = 
$$(k1 \times height [m]^3) + (k2 \times body weight [kg]) + k3$$

In this formula, k1 = 0.3669 for men and 0.3561 for women, k2 = 0.03219 for men and 0.03308 for women, and k3 = 0.6041 for men and 0.1833 for women

### Change in hemoglobin:

We will estimate the loss of hemoglobin (Hb) according to the formula:

### CONFIDENTIAL

Study number: S20-01617 Page 12 Version: 1.0 dated 05/05/2022

$$Hb_{loss} = blood\ volume\ x\ (Hb_i - Hb_e)\ x\ 0.001\ +\ Hb_t.$$

In this formula,  $Hb_{loss}(g) = the$  amount of hemoglobin lost through postoperative day 1,  $Hb_i(g/L) = the$  hemoglobin concentration preop,  $Hb_e(g/L) = the$  hemoglobin concentration on postoperative day 1, and  $Hb_t(g/L) = the$  amount of hemoglobin transfused.

The volume of total perioperative blood loss will be determined according to the following formula:

Total blood loss (ml) = 
$$1000 x \frac{Hb_{loss}}{Hb_i}$$

### Transfusion Criteria

All post op transfusions will be based on the recommendations from the American Association of Blood Banks to help reduce investigator bias secondary to unblinded staff. (Fillingham, Carson) Patients will only receive a blood transfusion under the following circumstances

- 1. Patient Hgb is less than 7g/dl or symptomatic and not responsive to IV fluid hydration
- 2. Patient has a history of cardiac disease and Hgb is less than 8g/dl or symptomatic and not responsive to IV fluid hydration

Patient has an active arterial thromboemebolic event or sepsis and Hgb is less than 10g/dl or symptomatic and not responsive to IV fluid hydration.

Study number: S20-01617 Version: 1.0 dated 05/05/2022

### 3.2 Schematic of Study Design

Enrollment

82 subjects: Obtain informed consent. Screen potential subjects by inclusion and exclusion criteria; obtain history, PreOP Hgb

### Randomize



### **GROUP 1**

IV TXA (2 doses) 2 grams of TXA 41 Subjects





### **GROUP 2**

Control Group No TXA 41 Subjects



**Post- OP** 

Surgical drain output, calculated total blood loss Hematoma formation, Need for transfusion


#### 4 **Study Enrollment and Withdrawal**

The researchers will approach patients scheduled for revision total shoulder arthroplasty who are eligible for participation in the study. Anesthesiology attendings fellows listed on the study team as well as other authorized researchers on the study team will consent and enroll patients pre-operatively.

#### 4.1 **Inclusion Criteria**

- 1. Patients older than 18 years old
- Patients younger than 90 years old 2.
- 3. Patients undergoing scheduled revision total shoulder arthroplasty
- 4. Patients who consent to be randomized

#### 4.2 **Exclusion Criteria**

- 1. Patients younger than 18
- 2. Patients older than 90 years old
- 3. Patients who are pregnant or breast-feeding women
- 4. Patients who are allergic to tranexamic acid
- 5. Patients with proximal humerus fracture or fracture sequelae
- 6. Patients who use estrogen containing medications (i.e. oral contraceptive pills)
- 7. Patients who have acquired disturbances of color vision
- 8. Patients with a history of any of the following diagnosis: `
  - Subarachnoid hemorrhage
  - o Active intravascular clotting
  - o Severe pulmonary disease (FEV <50% normal)
  - Plasma creatinine > 115 μmol/L in males, > 100 μmol/L in females, or hepatic failure)
  - (Renal impairment serum creatinine > 1.5 times the upper limit of normal NYU)
  - Preoperative anemia [Hemoglobin (Hb) < 11g/dL in females, Hb < 12 g/dL in males]
- 9. Patients who refuse blood products
- Patients undergoing hormone replacement therapy 10.
- 11. Patients with diagnosed or self-reported cognitive dysfunction;
- 12. Patients who are unable to understand or follow instructions;
- 13. Patients with severe liver disease, renal insufficiency, congestive heart failure, and/or significant heart disease:
- Patients with BMI over 50 14.
- 15. Any patient that the investigators feel cannot comply with all study related procedures.

#### 4.3 **Vulnerable Subjects**

No vulnerable populations will be enrolled in this study.

#### 4.4 **Recruitment and Consent**

This study will utilize EPIC to identify subjects and use the MCIT-managed HIPAA-compliant and encrypted version of Redcap in addition to the MCIT governed, firewall protected shared drive located on the NYU MCIT network, to manage and store relevant data.

### **Process of Consent**


During the subject's pre-surgical office visit, the study-surgeon will inform eligible patients about the study. Participants will be able to take a copy of the informed consent home to read through and take sufficient time to ask questions, discuss with family and/or research team prior to making an informed decision to participate on day of surgery. On day of surgery, informed consent will be obtained by a member of the research team after extensive discussion of risks and possible benefits of participation with the participants and their families. Consent forms will be IRB-approved and the participant will be asked to read and review the document. The presenter will explain the research study to the participant and answer any questions that may arise. All participants will receive a verbal explanation suited to their comprehension of the purposes, procedures, potential risks and their rights as research participants. Participants will have the opportunity to carefully review the written consent form and ask questions prior to signing. The participants will have the opportunity to discuss the study with their family or think about it prior to agreeing to participate. The participant will sign the informed consent document prior to any procedures being done specifically for the study. The participants may withdraw consent at any time throughout the course of the trial. A copy of the signed informed consent document will be offered to the participants for their records, a copy will be scanned into the subject's EMR, and the research staff will maintain a copy. The rights and welfare of the participants will be protected by emphasizing that the quality of their medical care will not be adversely affected if they decline to participate in this study.

A copy of the signed informed consent document will be offered to the patient, placed in the patient's electronic medical record and the original copy will be stored in the research regulatory binder. Any alteration to the standard consent process (e.g. use of an interpreter, consent document presented orally, etc.) and the justification for such alteration will likewise be documented.

### **Subject Capacity**

All subjects will be assessed for capacity to give informed consent by the anesthesiologist and the surgeon on the day of surgery. Capacity will be assessed through the subjects' ability to express understanding of the information presented to them, their ability to express a choice, their appreciation of how the study is relevant to them, and reasoning about how the study might impact them and others. Persons lacking capacity to consent will not be enrolled into the study.

If a subject requests information regarding opting out of further recruitment for all research, subjects will be directed to contact the PI, Dr. Arthur Hertling at 212-598-6085.

#### 4.5 **Duration of Study Participation**

While the study will be open for 3 years after beginning enrollment, the actual length of a study subject's participation is up to **two weeks**, as this corresponds with the surgical follow up visit, where the studysurgeon determines if the patient developed a post op hematoma.

#### 4.6 **Total Number of Participants and Sites**

In order to assess the superiority of the group receiving 2 g of TXA compared to control, we consulted the literature. In Vara (2017), in 102 patients, we determined that the mean calculated total blood loss was 1122.4 mL with a standard deviation of 411.6 in the TXA group vs. 1472.6 +/- 475.4 in the control group. Using the power equation with a SD of 444.6, an alpha of 0.05 and a power of 0.9, we estimate that 34 patients will be needed per group. Accounting for a possible attrition of up to 20%, we will aim to recruit 41 patients per group, or a total of 82 patients.

There is a single location for enrollment, NYU Langone Orthopedic Hospital.


#### 4.7 **Participant Withdrawal or Termination**

Participants are free to withdraw from participation in the study at any time upon request. An investigator may terminate participation in the study if:

- Any clinical adverse event (AE), laboratory abnormality, or other medical condition or situation occurs such that continued participation in the study would not be in the best interest of the participant
- The participant meets an exclusion criterion (either newly developed or not previously recognized) that precludes further study participation

#### 4.8 **Premature Termination or Suspension of Study**

This study may be temporarily suspended or prematurely terminated if there is sufficient reasonable cause. If the study is prematurely terminated or suspended, the PI will promptly inform the IRB and will provide the reason(s) for the termination or suspension.

Circumstances that may warrant termination or suspension include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to participants; 1.
- 2. Insufficient compliance to protocol requirements;
- 3. Data that are not sufficiently complete and/or evaluable

#### 5 **Risks and Benefits**

#### 5.1 **Potential Risks**

### Medication:

Risks of Intravenous TXA.

TXA works by preventing the breakdown of fibrin so there is a theoretical risk of thromboembolic events such as VTE, PE, MI with vascular stents, cerebral vascular occluisve disease. In patients using hormonal contraception, there is an increased risk of developing thromboembolic adverse reactions. TXA can cause visual disturbances. There is also a risk of seizures after TXA administration. Lastly, TXA can cause hypersentivity reactions.

### Risk of withholding TXA

Patients in the control arm of the study, will not NOT receive TXA. We do not believe this will increase bleeding risk for the control group as our NYU shoulder surgeons are nationally recognized experts in shoulder replacement surgery. Although studies have shown TXA decreases blood loss in this type of surgery, our shoulder surgeons believe it may not make a significant difference in total blood loss since the expected blood loss for this procedure at our institution is lower than in published studies. We attribute the lower blood loss in TSA surgery at our institution to the expertise of our surgeons. At NYU, due to the high clinical volume and expertise of the surgical team, all co -morbidities including blood loss is lower than published data. Therefore, we believe that TXA does not have to included as a routine prophylaxis. Although we have been providing TXA to all patients out of an abundance of caution, there is no data to clearly support the cost and potential risks of TXA is justified at our institution.

Study number: S20-01617 Page 17 Version: 1.0 dated 05/05/2022

### **Potential Benefits**

It is possible that study subjects who receive IV TXA may experience reduced incidence of hematoma, blood loss and blood transfusion during the study. It is also possible that subjects may not get any benefit from being in this research study. The study will help us optimize the TXA treatment protocol for future patients including discontinuing TXA use in total shoulder arthroplasy surgery. The knowledge gained from doing this study may benefit other patients in the future.

### 6 Statistical Analysis

### 6.1 General Approach

<u>Intention-to-treat</u>. The primary analysis will follow the intention-to-treat (ITT) principle in order to evaluate the true outcome of the intervention as experienced by the patient who is blinded to the intervention.

<u>Missing Data</u>. It is anticipated that the data for some subjects will be incomplete for various reasons: incorrect or missing data collection from OR nurse or floor nurses. All occurrences of incomplete data will be investigated to carefully document the reasons for the missing data. If the primary outcome, post op hemoglobin, surgical drain output cannot be ascertained with a reasonable degree of certainty, the patient will be excluded from the study.

# 6.2 Analysis of Endpoints

# **Primary Endpoints:**

- Calculated total blood loss (based on the change in pre-operative to POD 1 hemoglobin levels)
  - o Sub analysis of procedure depending on the type of surgical revision
- Surgical drain output (0-24 hours post op )

### **Secondary Endpoints:**

- Formation of Hematoma (At 2 week follow up visit. YES or NO)
- Need for Post op blood transfusion
- Operative time
- Development of adverse events, MI, PE, DVT

Data sub-analysis will be performed based on type of revision

- 1. Revision involving change of modular components (humeral head/glenosphere): **standard blood loss**
- 2. Revision involving removal and replacement of well fixed humerus component and/or glenoid component- high blood loss
- 3. Revision for infection that involves one or two stage process: moderate blood loss

All endpoints will be evaluated as fits the data set with graphical figures such as scatter plots, box-and-whisker plots, and frequency histograms to visualize the distribution of these outcomes and their relationships to covariates and treatment assignment. When appropriate descriptive graphical and tabular methods will also be estimated and presented in a graphical figure.


### **6.2.1** Baseline Descriptive Statistics

The following patient data will be recorded: age, gender, height, weight, date of admission, date of discharge, laterality, surgical approach, implants used, duration of surgery, contamination, ASA, comorbidities (smoking, cardiac history, diabetes etc.), CBC (WBC, PCV, HGB, RBC, indices, platelet count, differential), and medications. All of this information will be accessible in the patient's medical record. Descriptive statistics will be used to summarize variables with mean and standard deviation for continuous variables, or percentages for categorical variables.

### Sample Size:

Power analysis was performed for the primary outcome of total blood loss (See 4.6).

The primary outcome of total blood loss will be tested using two one sided t-tests (TOST) for equivalence testing between intervention groups whereby a p-value of <0.05 represents statistical equivalence. Additionally, demographical and baseline comparisons between intervention groups will be made usisng an analysis os variance (ANOVA) for continuous measurements or a chi-squared or Fischer's exact test for categorical variables. Significance will be set at a p-value of <0.05

### 6.3 Enrollment/Randomization/Masking Procedures

We will utilize a simple-randomization method to create two equal groups of subjects as mentioned in the schematic study design (3.2). Additionally, we will use a computer software, randomization.com, to generate the randomization assignment for all participants. Someone that is not a stakeholder in the study will make randomization opaque envelopes, which includes the study ID number, the treatment assignment, and dosage specifics. These randomization envelopes will then be distributed to the anesthesiologist pre-operatively by the authorized researcher after informed consent is obtained.

### 6.4 Breaking the Study Blind/Participant Code

If there is any adverse event related to the drug, we will break the blind for the subject and randomization will be disclosed to the patient.

### 7 Assessment of Safety

An **adverse event** (AE) is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. Intercurrent illnesses or injuries should be regarded as adverse events. Abnormal results of diagnostic procedures are considered to be adverse events if the abnormality:

- results in study withdrawal
- is associated with a serious adverse event
- is associated with clinical signs or symptoms
- leads to additional treatment or to further diagnostic tests
- is considered by the investigator to be of clinical significance

### 7.1 Definition of Serious Adverse Events (SAE)

### **Serious Adverse Event**

Adverse events are classified as serious or non-serious. A serious adverse event is any AE that is:

- fatal
- life-threatening
- requires or prolongs hospital stay

### CONFIDENTIAL

Study number: S20-01617 Page 19 Version: 1.0 dated 05/05/2022

results in persistent or significant disability or incapacity

- a congenital anomaly or birth defect
- an important medical event

Important medical events are those that may not be immediately life threatening, but are clearly of major clinical significance. They may jeopardize the subject, and may require intervention to prevent one of the other serious outcomes noted above. For example, drug overdose or abuse, a seizure that did not result in in-patient hospitalization or intensive treatment of bronchospasm in an emergency department would typically be considered serious.

All adverse events that do not meet any of the criteria for serious will be regarded as **non-serious adverse events**.

### 7.2 Classification of an Adverse Event

### 7.2.1 Severity of Event

For AEs not included in the protocol defined grading system, the following guidelines will be used to describe severity.

- 1. **Mild** Events require minimal or no treatment and do not interfere with the participant's daily activities.
- 2. **Moderate** Events result in a low level of inconvenience or concern with the therapeutic measures. Moderate events may cause some interference with functioning.
- 3. **Severe** Events interrupt a participant's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually potentially life-threatening or incapacitating.

### 7.2.2 Relationship to Study Agent

The clinician's assessment of an AE's relationship to study agent (drug, biologic, device) is part of the documentation process, but it is not a factor in determining what is or is not reported in the study. If there is any doubt as to whether a clinical observation is an AE, the event will be reported. All AEs must have their relationship to study agent assessed. For all collected AEs, the clinician who examines and evaluates the participant will determine the AE's causality based on temporal relationship and his/her clinical judgment. The degree of certainty about causality will be graded using the categories below.

- 1. **Definitely Related** There is clear evidence to suggest a causal relationship, and other possible contributing factors can be ruled out. The clinical event, including an abnormal laboratory test result, occurs in a plausible time relationship to drug administration and cannot be explained by concurrent disease or other drugs or chemicals.
- 2. **Probably Related** There is evidence to suggest a causal relationship, and the influence of other factors is unlikely. The clinical event, including an abnormal laboratory test result, occurs within a reasonable time after administration of the drug, is unlikely to be attributed to concurrent disease or other drugs or chemicals, and follows a clinically reasonable response on withdrawal).
- 3. **Possibly Related** There is some evidence to suggest a causal relationship (e.g., the event occurred within a reasonable time after administration of the trial medication). However, other factors may have contributed to the event (e.g., the participant's clinical condition, other concomitant events). Although an AE may rate only as "possibly related" soon after discovery, it can be flagged as requiring more information and later be upgraded to "probably related" or "definitely related," as appropriate.
- 4. **Unlikely to be related** A clinical event, including an abnormal laboratory test result, whose temporal relationship to drug administration makes a causal relationship improbable (e.g., the event did not CONFIDENTIAL

Study number: S20-01617 Page 20 Version: 1.0 dated 05/05/2022

occur within a reasonable time after administration of the trial medication) and in which other drugs or chemicals or underlying disease provides plausible explanations (e.g., the participant's clinical condition, other concomitant treatments).

5. **Not Related** – The AE is completely independent of study drug administration, and/or evidence exists that the event is definitely related to another etiology. There must be an alternative, definitive etiology documented by the clinician.

Dr. Arthur Hertling will be responsible for determining whether an AE is expected or unexpected. An AE will be considered unexpected if the nature, severity, or frequency of the event is not consistent with the risk information previously described for the study agent.

# 7.3 Time Period and Frequency for Event Assessment and Follow-Up

The occurrence of an AE or SAE may come to the attention of study personnel during study visits and interviews of a study participant presenting for medical care, or upon review by a study monitor. All AEs including local and systemic reactions not meeting the criteria for SAEs will be captured on the appropriate RF. Information to be collected includes event description, time of onset, clinician's assessment of severity, relationship to study product (assessed only by those with the training and authority to make a diagnosis), and time of resolution/stabilization of the event. All AEs occurring while on study must be documented appropriately regardless of relationship. All AEs will be followed to adequate resolution.

Any medical condition that is present at the time that the participant is screened will be considered as baseline and not reported as an AE. However, if the study participant's condition deteriorates at any time during the study, it will be recorded as an AE. UPs will be recorded in the data collection system throughout the study.

Changes in the severity of an AE will be documented to allow an assessment of the duration of the event at each level of severity to be performed. AEs characterized as intermittent require documentation of onset and duration of each episode.

The PI will record all reportable events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. At each study visit, the investigator will inquire about the occurrence of AE/SAEs since the last visit. Events will be followed for outcome information until resolution or stabilization. As per NYU IRB policy, we will abide by the time frame for reporting AE/SAE's. The time frame for reporting SAE and UP to the DSMB is by telephone within 24 hours of awareness of the event. The time frame for reporting SAE and UP to the IRB is to submit reports promptly but no later than 5 working days from the time the investigator becomes aware of the event.

All unresolved adverse events will be followed by the investigator until the events are resolved, the subject is lost to follow-up, or the adverse event is otherwise explained. At the last scheduled visit, the investigator will instruct each subject to report any subsequent event(s) that the subject, or the subject's personal physician, believes might reasonably be related to participation in this study. The investigator will notify the medical center IRB of any death or adverse event occurring at any time after a subject has discontinued or terminated study participation that may reasonably be related to this study. The medical center IRB will also be notified if the investigator should become aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a subject that has participated in this study.


#### 7.4 **Safety Oversight**

It is the responsibility of the Principal Investigator to oversee the safety of the study at his/her site. This safety monitoring will include careful assessment and appropriate reporting of adverse events as noted above, as well as the construction and implementation of a site data and safety-monitoring plan. Medical monitoring will include a regular assessment of the number and type of serious adverse events. Additionally, the study will have a DSMB.

The DSMB will be made up of the Principal Investigator, Arthur Hertling M.D. and Co-investigator. Young Kwon M.D. All members of the DSMB are board certified physicians in their respective specialties Anesthesiology and Orthopedic Surgery.

The DSMB will review safety data after the first five enrolled subjects and every three months thereafter. All unanticipated problems that increase risk to the subjects will be reported to the IRB per NYUSOM IRB policy.

During these meetings, the DSMB will review and analyze any unanticipated problems or adverse events involving risk to the patient including thromboembolic events such as VTE, PE, MI with vascular stents, cerebral vascular occluisve disease.

Specific study stopping points is the occurrence of a serious adverse event such as a severe allergic reaction to TXA. Additionally, after 5 patients in each group have completed all study related procedures, a brief safety analysis will be done by the Principal Investigator, Arthur Hertling M.D. Events will be reported to the anesthesia department QA.

Additionally, the DSMB will perform an interim safety and data analysis after 40 patients have completed all study related visits. Outcomes of these reviews will be submitted to the IRB in an annual progress report at the time of Continuing Review.

#### 8 **Source Documents and Access to Source Data/Documents**

Source data is all information, original records of clinical findings, observations, or other activities in a clinical trial necessary for the reconstruction and evaluation of the trial. Source data are contained in source documents. Examples of these original documents, and data records include: hospital records, clinical and office charts, laboratory notes, memoranda, subjects' diaries or evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies or transcriptions certified after verification as being accurate and complete, microfiches, photographic negatives, microfilm or magnetic media, x-rays, subject files, and records kept at the pharmacy, at the laboratories, and at medicotechnical departments involved in the clinical trial.

The study case report form (CRF) is the primary data collection instrument for the study. All data requested on the CRF must be recorded. All missing data must be explained. If a space on the CRF is left blank because the procedure was not done or the question was not asked, write "N/D". If the item is not applicable to the individual case, write "N/A". All entries will be printed legibly in black ink.

Access to study records will be limited to IRB-approved members of the study team. The investigator will permit study-related monitoring, audits, and inspections by the IRB/EC, the sponsor, government regulatory bodies, and University compliance and quality assurance groups of all study related documents


(e.g. source documents, regulatory documents, data collection instruments, study data etc.). The investigator will ensure the capability for inspections of applicable study-related facilities (e.g. pharmacy, diagnostic laboratory, etc.).

### 9 Ethics/Protection of Human Subjects

### 9.1 Ethical Standard

The investigator will ensure that this study is conducted in full conformity with Regulations for the Protection of Human Subjects of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, and/or the ICH E6.

### 9.2 Institutional Review Board

The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the IRB for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. All changes to the consent form will be IRB approved; a determination will be made regarding whether previously consented participants need to be re-consented.

### 9.3 Participant and Data Confidentiality

Participant confidentiality is strictly held in trust by the participating investigators, their staff, and the sponsor(s) and their agents. Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study or the data will be released to any unauthorized third party without prior written approval of the sponsor.

The study monitor, representatives of the IRB may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the participants in this study. The clinical study site will permit access to such records.

The study participant's contact information will be securely stored at each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by local IRB and Institutional regulations.

Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at NYU Langone Medical Center. This will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management system (REDCap) used by the clinical site and by NYU Langone Medical Center research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and archived at the NYU Langone Medical Center.

Study number: S20-01617 Page 23 Version: 1.0 dated 05/05/2022

# 10 Data Handling and Record Keeping

### 10.1 Data Collection and Management Responsibilities

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site PI. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data. Black ink is required to ensure clarity of reproduced copies. When making changes or corrections, cross out the original entry with a single line, and initial and date the change. DO NOT ERASE, OVERWRITE, OR USE CORRECTION FLUID OR TAPE ON THE ORIGINAL.

Copies of the electronic CRF (eCRF) will be provided for use as source documents and maintained for recording data for each participant enrolled in the study. Data reported in the eCRF derived from source documents should be consistent with the source documents or the discrepancies should be explained and captured in a progress note and maintained in the participant's official electronic study record.

Clinical data (including AEs, concomitant medications, and expected adverse reactions data) and clinical laboratory data will be entered into Redcap. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate. Clinical data will be entered directly from the source documents.

### 10.2 Study Records Retention

Study documents will be retained for the longer of 3 years after close-out, 5 years after final reporting/publication, or 2 years after the last approval of a marketing application is approved for the drug for the indication for which it is being investigated or 2 years after the investigation is discontinued and FDA is notified if no application is to be filed or if the application has not been approved for such indication. No records will be destroyed without the written consent of the sponsor, if applicable. It is the responsibility of the sponsor to inform the investigator when these documents no longer need to be retained.

### 10.3 Protocol Deviations

It is the responsibility of the site PI/study staff to use continuous vigilance to identify and report deviations within 7 working days of identification of the protocol deviation, or within 7 working days of the scheduled protocol-required activity.

Protocol deviations will be reported to the local IRB per their guidelines. The site PI/study staff is responsible for knowing and adhering to their IRB requirements.

### 10.4 Publication and Data Sharing Policy

This trial will be registered with the clinicaltrials.gov as per the ICMJE policy, and the Section 801 of the Food and Drug Administration Amendments Act of 2007.

Study number: S20-01617 Page 24 Version: 1.0 dated 05/05/2022

### 11 Study Finances

### 11.1 Funding Source

No funding source present.

### 11.2 Costs to the Participant

There are no expected costs to the subjects.

### 11.3 Participant Reimbursements or Payments

Participants will not receive any financial compensation for participation in this study.

### 12 Conflict of Interest Policy

The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the trial. The study leadership has established policies and procedures for all study group members to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest.

Any investigator who has a conflict of interest with this study (patent ownership, royalties, or financial gain greater than the minimum allowable by their institution, etc.) must have the conflict reviewed by the NYU Langone Conflict of Interest Management Unit (CIMU) with a Committee-sanctioned conflict management plan that has been reviewed and approved by the study sponsor prior to participation in this study. All NYULMC investigators will follow the applicable conflict of interest policies.

Study number: S20-01617 Page 25 Version: 1.0 dated 05/05/2022

### 13 References

1. McCormack PL. Tranexamic acid. A Review of its use in the treatment of hyperfibrinolysis. Drug. 2012 Mar 26; 72 (5): 585-617

- 2. Budge M. Topical and intravenous tranexamic acid are equivalent in decreasing blood loss in total shoulder arthroplasty. Journal of Shoulder and Elbow Athroplasty. 2019. 3:1-5
- 3. Kirsch JM, Bedi A, Horner N, Wiater JM, Pauzenberger L, Koueiter DM, et al. Tranexamic acid in shoulder arthroplasty: a systematic review and meta-analysis. JBJS Rev. 2017;5(9):e3. doi: 10.2106/JBJS.RVW.17.00021
- 4. Dines, J S, Fealy, S, Strauss, E, Allen, A, Craig, EV, Warren, RF, Dines, DM. Outcomes Analysis of Revision Total Shoulder Replacement, JBJS: July 2006 Volume 88 Issue 7 p 1494-1500
- 5. Burns KA, Robbins LM, LeMarr AR, Childress AL, Morton DJ, Wilson ML. Estimated blood loss and anemia predict transfusion after total shoulder arthroplasty: a retrospective cohort study. *JSES Open Access*. 2019;3(4):311-315. Published 2019 Oct 15.
- 6. King JJ, Patrick MR, Schnetzer RE, et al. Multivariate Analysis of Blood Transfusion Rates After Shoulder Arthroplasty. *J Surg Orthop Adv.* 2017;26(1):40-47.
- 7. Saltzman, BM, Chalmers, PN, Gupta, Anil, Romeo, AA, Nicholson, GP. Complication rates comparing primary with revision reverse total shoulder arthroplasty. Journal of Shoulder and Elbow Surgery. Volume 23, Issue 11, 2014, 1647-1654,
- 8. Favard L. Revision of total shoulder arthroplasty. Orthopaedics & Traumatology: Surgery & Research, Volume 99, Issue 1, Supplement, 2013, Pages S12-S21,
- 9. Yang L, Du S, Sun Y. Is combined topical and intravenous tranexamic acid superior to single use of tranexamic acid in total joint arthroplasty?: A meta-analysis from randomized controlled trials. Medicine (Baltimore) 2017;96:e7609.
- 10. G.L. Cvetanovich, Y.A. Fillingham, M. O'Brien, B. Forsythe, B.J. Cole, N.N. Verma, et al. Tranexamic acid reduces blood loss after primary shoulder arthroplasty: a double-blind, placebo-controlled, prospective, randomized controlled trial. JSES Open Access, 2 (2018), pp. 23-27
- 11. Fillingham YA, Darrith B, Calkins TE, Abdel MP, Malkani AL, Schwarzkopf R, Padgett DE et al. 2019 Mark Coventry Award: A randomized clinical trial of tranexamic acid in revision total knee arthroplasty. Does the dosing regimen matter? The Bone and Joint Journal. 2019:101
- 12. Fillingham YA, Ramkumar DB, Jevsevar DS, Yates AJ, Bini SA, Clarke HD, Schemitsch E, Johnson RL, Memtsoudis SG, Sayeed SA, Sah AP, Della Valle CJ. Tranexamic Acid Use in Total Joint Arthroplasty: The Clinical Practice Guidelines Endorsed by the American Association of Hip and Knee Surgeons, American Society of Regional Anesthesia and Pain Medicine, American Academy of Orthopaedic Surgeons, Hip Society, and Knee Society. J Arthroplasty. 2018 Oct;33(10):3065-3069..
- 13. Abildgaard JT, McLemore R, Hattrup SJ. Tranexamic Acid decreases blood loss in total shoulder arthroplasty and reverse total shoulder arthroplasty. JSES. 2016; 25: 1643-1648 CONFIDENTIAL

Study number: S20-01617 Page 26 Version: 1.0 dated 05/05/2022

14. Gillespie R, Shishani Y, Joseph S et al. Neer Award 2015: A randomized prospective evaluation on the effectiveness of tranexamic acid in reducing blood loss after total shoulder arthroplasty. JSES. 2015; 24:1679-1684

- 15. Vara AD, Koueiter DM, Pinkas DE et al. Intravenous TXA reduces total blood loss in reverse total shoulder arthroplasty: a propspective double blind randomized trial. JSES. 2017; 26:1383-1389
- 16. Freidman RJ, Gordon E, Butler B et al. Tranexamic acid decreases blood loss after total shoulder arthroplasty. JSES. 2016; 25: 614-618
- 17. Tsukada S, Kurosaka K, Nishino M et al. Intraoperative Inatravenous and intra-articular plus postoperative intravenous tranexamic acid in total knee arthroplasty. JBJS. 2020; 102: 687-92
- 18. Carson JL, Grossman BJ, Kleinman S, et al. Red blood cell transfusion: a clinical practice guideline from the AABB\* Ann Intern Med 2012;157:49-58
- 19. Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32.

### **Attachments**

These documents are relevant to the protocol, but they are not considered part of the protocol. They are stored and modified separately. As such, modifications to these documents do not require protocol amendments.